CLINICAL TRIAL: NCT02479087
Title: IMMUNE TOLERANCE INDUCTION, BY FACTOR VIII CONCENTRATE CONTAINING VON WILLEBRAND FACTOR, IN SEVERE OR MODERATE HAEMOPHILIA A PATIENTS WITH INHIBITORS
Brief Title: Safety/Efficacy Study to Assess Whether FVIII/VWF Concentrate Can Induce Immune Tolerance in Haemophilia A Patients
Acronym: ITI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Sintesi Research Srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCG-CNS-001
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Hemophilia A
Keywords: von Willebrand Factor; Factor VIII; Hemorrhage; Immune Tolerance; Hemophilia A
MeSH Terms: conditions — Hemophilia A; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plasma-derived FVIII/VWF concentrate (Experimental): The drug will be delivered through intravenous slow infusion/injection. The starting dosage can vary between the minimum dosage of 50 IU/Kg 3 times a week up to a maximum of 200 IU/kg per day.
  This starting dosage will be decided by the Principal Investigator according to patient's condition and other variables.
  The initial dosage can be then adjusted on the base of response.
  Interventions: Drug: Plasma-derived FVIII/VWF concentrate

INTERVENTIONS:
Drug: Plasma-derived FVIII/VWF concentrate — The investigational treatment is with lyophilized plasma-derived Factor VIII. The product belongs to the factor VIII concentrates class, containing also VW Factor in an average ratio VW/VIII of > 1: 4.5.
  The product is as a powder and a solvent solution for continuous infusion of Factor VIII. The specific activity of Factor VIII is of approximately 80 IU/mg protein.
  The number of units of FVIII administered is expressed in International Units (IU), which are consistent with current WHO standards for products containing Factor VIII. The activity of Factor VIII in plasma is expressed either as a percentage (compared to normal human plasma) or in International Units (compared to the international standard for FVIII in plasma).
  Other Names: Emoclot

SUMMARY:
The purpose of this study is to assess the role of a FVIII/VWF complex concentrate (Emoclot) in successfully inducing immune tolerance (I.T.I.) in patients with Haemophilia A with inhibitors, including patients at high risk of failure.

DETAILED DESCRIPTION:
The development of factor VIII inhibitors occurs in approximately 30 to 40% of patients with severe Haemophilia A. The main negative clinical and cost consequence is the ineffectiveness of replacement therapy in patients with high-titer antibodies, who have a shorter life and greater morbidity than those who do not develop inhibitors. It is known from immunology that a regular and frequent exposure to the antigen of FVIII can induce tolerance of the immune system of the patient with inhibitors. This effect, called "immune tolerance induction" (ITI) is usually achieved after a prolonged exposure of the patient to FVIII, and is a common way of managing the condition of patients with inhibitors as well as the treatment of bleeding episodes with large amounts of hemostatic agents. In vitro and retrospective clinical studies suggest that FVIII/VWF complex concentrates may have less immunogenicity with respect to those plasma-derived concentrates purified with monoclonal antibodies (MABs), and recombinant DNA factor VIII concentrates (rFVIII), in both which the von Willebrand factor (VWF) is absent. Immune tolerance induction (ITI) showed to be effective in about 70% of Haemophiliacs with inhibitors. Poor prognosis factors have been identified by different registries: age ≥ 6 years, ITI started >1 year from inhibitor development, inhibitor peaks >200 BU, inhibitor titer >10 BU at the start of ITI and previously failed ITI. The results of clinical studies suggest that complex concentrates of VWF/FVIII can be effective in ITI, even in patients at high risk of failure. To explain these findings, a role for VWF (i.e. prolonged antigen exposure) has been hypothesized.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects (his/her parent/legal representative), must have given a written informed consent.
2. Male children: age <12 years.
3. Severe or moderate Haemophilia A (FVIII <2%).
4. High responders (clinical history of inhibitor peak > 5BU) or low-responders (clinical history of inhibitor peak < 5 BU) with potential bleedings, assessed by responsible physicians as not to be treated with high FVIII doses.
5. Any level of inhibitor at study enrollment.
6. Willingness and ability to participate in the study.
7. No other experimental treatments (involving or not FVIII concentrates).

Exclusion Criteria:

1. Any clinically relevant abnormality, in hematological, biochemical and urinary routine examinations, or any condition or treatment which in the investigator's opinion, makes the patient not eligible for the study.
2. Intolerance to active substances or to any of the excipients of FVIII / VWF concentrates.
3. Concomitant systemic treatment with immunosuppressive drugs.

Max Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy: evaluation of the success of IT induction | Up to33 months
  Success:Inhibitor disappearance/reduction to <0.6 BU/ml with FVIII activity recovery of at least ≥ 66% within 33 months of treatment ; Partial Success: inhibitor reduction to <5 BU/ml with clinical response to FVIII treatment, not followed by an inhibitor increase to values >5 BU/ml for a treatment period of 6 months on demand, or for 12 months of prophylactic treatment; No Response (Failure):Failure in relation to the above criteria defining complete response and partial response within 33 months, OR a reduction of the concentration of the inhibitor, less than 20%, compared to the peak of inhibitor in the IT, in every period of 6 months after the first 3 months of treatment. This implies that 9 months represents the minimum period of treatment and 33 months the maximum possible duration of ITI without success, OR patient withdrawal from the study for any reason.

SECONDARY OUTCOMES:
Safety (adverse events) | Up to 33 months
  Description and incidence of adverse events during the course of prophylactic treatment, with severity, correlation with the investigational product and final outcome.
Analysis of treatment compliance | Up to 33 months
  Description of the patient's adherence to the optimal prolonged treatment.
Efficacy evaluation - Time to achieve ITI | Up to 33 months
  Time to achieve the complete or partial response (as defined in the primary outcome measure).
Evaluation of the cost of therapy | Up to 33 months
  Recording of overall amount of direct costs of therapy.
Efficacy evaluation - IT persistence | Up to 33 months+ 12 months FU
  Absence of relapse, assessed at 12 months from IT achievement
Efficacy evaluation - FVIII genetic defect role in IT achievement | Up to 33 months
  Role of FVIII mutations in influencing IT achievement
Efficacy evaluation - Role of an immediate IT to delayed IT in IT induction. | Up to 33 months
  Time elapsing between the onset of the inhibitor and the beginning of treatment and its importance for induction of IT in achieving primary endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Pier Mannuccio Mannucci, MD, Study Chair — IRCCS Fondazione Ca' Granda Ospedale Maggiore Policlinico; Flora Peyvandi, MD, Study Director — Università di Milano, IRCCS Fondazione Ca' Granda Ospedale Maggiore Policlinico; Elena Santagostino, MD, Study Director — Centro Emofilia e Trombosi Angela Bianchi Bonomi, IRCCS Fondazione Ospedale Maggiore Policlinico
Locations (4):
- Egypt (2):
  - Ain Shams Pediatric hospital, Ain Shams University, Cairo
  - Almoneera Pediatric Cairo University Hospital (Abu El- Reesh), Cairo
- India (2):
  - St. John's Medical College Hospital, Bangalore
  - All India Institute of Medical Sciences, New Delhi

REFERENCES:
- [Background] Gilles JG, Saint-Remy JMR. Recombinant and plasma-derived factor VIII are immunologically distinct in in vitro assays. Thromb Haemost 1995; 73:1213.
- [Background] Guerois C, Laurian Y, Rothschild C, Parquet-Gernez A, Duclos AM, Negrier C, Vicariot M, Fimbel B, Fressinaud E, Fiks-Sigaud M, et al. Incidence of factor VIII inhibitor development in severe hemophilia A patients treated only with one brand of highly purified plasma-derived concentrate. Thromb Haemost. 1995 Feb;73(2):215-8. PMID 7792732
- [Background] Yee TT, Williams MD, Hill FG, Lee CA, Pasi KJ. Absence of inhibitors in previously untreated patients with severe haemophilia A after exposure to a single intermediate purity factor VIII product. Thromb Haemost. 1997 Sep;78(3):1027-9. PMID 9308748
- [Background] Teitel JM. Safety of coagulation factor concentrates. Haemophilia. 1998 Jul;4(4):393-401. doi: 10.1046/j.1365-2516.1998.440393.x. PMID 9873760
- [Background] Rokicka-Milewska R, Klukowska A, Dreger B, Beer H-J. Incidence of factor VIII inhibitor development in previously untreated Haemophilia A patients after exposure to a double viral inactivated factor VIII concentrate. Ann Hematol 1999; 78 (suppl 1)
- [Background] Aznar JA, Lorenzo JI, Molina R, Haya S, Querol F, Dasi MA. Zero incidence of inhibitor development in previously treated haemophilia A, HIV-negative patients upon exposure to a plasma-derived high-purity and double viral inactivated factor VIII concentrate. Haemophilia. 1998 Jan;4(1):21-4. doi: 10.1046/j.1365-2516.1998.00139.x. PMID 9873861
- [Background] Smith MP, Rice KM, Savidge GF. Successful clinical use of a plasma-derived, dual virus inactivated factor VII concentrate incorporating solvent-detergent and dry heat treatment. Thromb Haemost. 1997 Feb;77(2):406-7. No abstract available. PMID 9157608
- [Background] Sukhu K, Keeling DM, Giangrande PL. Variation in inhibitor reactivity in acquired haemophilia A with different concentrates. Clin Lab Haematol. 2000 Oct;22(5):287-90. doi: 10.1046/j.1365-2257.2000.00328.x. PMID 11122270
- [Background] Gensana M, Altisent C. Aznar JA, Casana P, Hernandez F, Jorquera JI, Magallon M, Massot M, Puig L. Factor VIII inhibitors directed to the A2 domain and the light chain may also show less reactivity to FVIII complexed with VWF. World Federation of Haemophilia, The Hague, May 1998, (Abstract book).
- [Background] Suzuki T, Arai M, Amano K, Kagawa K, Fukutake K. Factor VIII inhibitor antibodies with C2 domain specificity are less inhibitory to factor VIII complexed with von Willebrand factor. Thromb Haemost. 1996 Nov;76(5):749-54. PMID 8950785
- [Background] Gensana M, Altisent C, Aznar JA, Casana P, Hernandez F, Jorquera JI, Magallon M, Massot M, Puig L. Influence of von Willebrand factor on the reactivity of human factor VIII inhibitors with factor VIII. Haemophilia. 2001 Jul;7(4):369-74. doi: 10.1046/j.1365-2516.2001.00526.x. PMID 11442641
- [Background] Berntorp E, Ekman M, Gunnarsson M, Nilsson IM. Variation in factor VIII inhibitor reactivity with different commercial factor VIII preparations. Haemophilia. 1996 Apr;2(2):95-9. doi: 10.1111/j.1365-2516.1996.tb00022.x. PMID 27214015
- [Background] Kreutz W: Immune tolerance induction (ITI) in Haemophilia A-patients with inhibitors - the choice of concentrate affecting success. Haematologica 2001; 86 (S4):16-20
- [Background] Kreuz W, Steiner J, Auerswald G, Beeg T, Becker S. Successful immunetolerance therapy of FVIII-inhibitor in chldren after changing from high to intermediate purity FVIII concentrate. Ann Hematol 1996; 72 (suppl 1).
- [Background] Orsini F, Rotschild C, Beurrier P, Faradji A, Goudemand J, Polack B. Immune tolerance induction with highly purified plasma-derived factor VIII containing von Willebrand factor in hemophilia A patients with high-responding inhibitors. Haematologica. 2005 Sep;90(9):1288-90. PMID 16154861
- [Background] Gringeri A, Musso R, Mazzucconi MG, Piseddu G, Schiavoni M, Pignoloni P, Mannucci PM; RITS-FITNHES Study Group. Immune tolerance induction with a high purity von Willebrand factor/VIII complex concentrate in haemophilia A patients with inhibitors at high risk of a poor response. Haemophilia. 2007 Jul;13(4):373-9. doi: 10.1111/j.1365-2516.2007.01484.x. PMID 17610550
- [Background] Mauser-Bunschoten EP, Nieuwenhuis HK, Roosendaal G, van den Berg HM. Low-dose immune tolerance induction in hemophilia A patients with inhibitors. Blood. 1995 Aug 1;86(3):983-8. PMID 7620189
- [Background] Hay CR, DiMichele DM; International Immune Tolerance Study. The principal results of the International Immune Tolerance Study: a randomized dose comparison. Blood. 2012 Feb 9;119(6):1335-44. doi: 10.1182/blood-2011-08-369132. Epub 2011 Nov 18. PMID 22101900
- [Background] Haya S, Casaña P, Moret A, Cid RA, Cabrera N, Abad L, Aznar AJ. Immunotolerance Induction Treatments in Hemophilia. J.of Coagulation Disorders 2009; 1(1): 37-42.
- [Background] Colowick AB, Bohn RL, Avorn J, Ewenstein BM. Immune tolerance induction in hemophilia patients with inhibitors: costly can be cheaper. Blood. 2000 Sep 1;96(5):1698-702. PMID 10961866
- [Background] Coppola A, Di Minno MN, Santagostino E. Optimizing management of immune tolerance induction in patients with severe haemophilia A and inhibitors: towards evidence-based approaches. Br J Haematol. 2010 Sep;150(5):515-28. doi: 10.1111/j.1365-2141.2010.08263.x. Epub 2010 Jun 22. PMID 20573153